CLINICAL TRIAL: NCT00303134
Title: Human Islet Cell Transplantation in Type 1 Diabetic Patients
Brief Title: Islet Cell Transplants for Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: poor intermediate-term results
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0105004956
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: islet cell; diabetes; transplant; immunosuppression; autoimmunity; alloimmunity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases | interventions — Islets of Langerhans Transplantation

ARMS (1):
- Islet Cell Transplantation (Experimental)
  Interventions: Drug: Islet Cell Transplantation

INTERVENTIONS:
Drug: Islet Cell Transplantation — Islet Cell Transplantation for patients with type 1 diabetes mellitus

SUMMARY:
The purpose of this study is to test the safety and efficacy of islet cell transplants for the treatment of type 1 diabetes mellitus. It has been shown that normal control of blood sugar levels can prevent progression of complications (such as kidney disease, nerve damage, and vascular disease) from diabetes. This research study is designed to see if normal blood sugar control can be achieved by transplanting pancreatic islet cells into your liver, which may reduce or eliminate your need for insulin. Patients may qualify to participate in this research study if they have type 1 diabetes mellitus for at least five years and meet at least one of the following criteria:

* Experience hypoglycemic unawareness - Defined as inability to tell when blood glucose is low (for example, may not feel symptoms such as shaking, sweating, and rapid heartbeat that usually signify that glucose is low)
* Have been hospitalized several times in the past year for low blood sugar and/or high blood sugar
* Have complications of diabetes such as retinopathy, kidney problems, or neuropathy

ELIGIBILITY:
Inclusion Criteria:

- Enrolling subjects must have Type 1 diabetes mellitus for more than 5 years, complicated by at least one of the following situations that persist despite intensive insulin management efforts. (Intensive management is defined as monitoring of glucose values at home no less than three times each day and by the administration of three or more insulin injections each day. Such management must be monitored in close cooperation with an endocrinologist or primary care physician, as defined by at least three contacts during the previous 12 months. If an endocrinologist did not participate in the ongoing management effort during the past year, then an independent endocrinologist must assess the adequacy of the management efforts prior to enrollment.) The complicating situations are:

a. Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels of < 54 mg/dL, b. Metabolic lability/instability, characterized by two or more episodes of severe hypoglycemia and which is associated with a blood glucose below 54 mg/dl OR two or more hospital visits for diabetic ketoacidosis over the last year, c. Despite efforts at optimal glucose control, progressive secondary complications of diabetes as defined by: i) Retinopathy-a minimum of a three step progression using the Early Treatment Diabetic Retinopathy Study (ETDRS) grading system 44,or an equivalent progression as certified by an ophthalmologist familiar with diabetic retinopathy, or ii) Nephropathy-a confirmed rise of 50 µg/min (72 mg/24h) of microalbuminuria or greater over at least three months (beginning anytime within the past two years) despite the use of an ACE inhibitor, or iii) Neuropathy-persistent or progressing autonomic neuropathy (gastroparesis, postural hypotension, neuropathic bowel or bladder) or persistent or progressing severe peripheral painful neuropathy not responding to usual management (e.g., tricyclics, gabapentin, or carbamazepine).

Exclusion Criteria:

1. Severe co-existing cardiac disease, characterized by any one of these conditions:

   * Recent myocardial infarction (within past six months), or
   * Angiographic evidence of non-correctable coronary artery disease, or
   * Evidence of ischemia on functional cardiac exam (functional testing is required for all subjects, with a stress echo test recommended for subjects with a history of ischemic disease). Patients unable to perform an exercise stress echocardiogram test will undergo adenosine vasodilator stress test, and if there is a history of bronchospasm, will undergo dobutamine stress test.
2. Active alcohol or substance abuse-includes cigarette smoking (must be abstinent for six months). Active alcohol abuse should be considered using the current NIAAA definitions, whereby alcohol abuse is defined by a pattern of drinking that is accompanied by one or more of the following situations within a 12-month period:

   * Failure to fulfill major work, school, or home responsibilities;
   * Drinking in situations that are physically dangerous, such as while driving a car or operating machinery;
   * Recurring alcohol-related legal problems, such as being arrested for driving under the influence of alcohol or for physically hurting someone while drunk;
   * Continued drinking despite having ongoing relationship problems that are caused or worsened by the effects of alcohol.
3. Psychiatric disorder making the subject not a suitable candidate for transplantation, e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication. (A psychological or psychiatric consultation is required only if considered necessary by some current indication or history.)
4. History of non-adherence to prescribed regimens
5. Active infection including hepatitis C, hepatitis B, HIV, or TB (or under treatment for suspected TB)
6. Any history of or current malignancies except squamous or basal skin cancer
7. BMI > 26 kg/m2
8. C-peptide response to arginine stimulation (5 gm I.V.) (any C-peptide ≥ 0.3 ng/mL at 2, 3, 4, 5, 7 and 10 min post-infusion)
9. Inability to provide informed consent
10. Age less than 18 or greater than 65 years
11. Creatinine clearance <80 mL/min/1.73 m2
12. Serum creatinine >1.6 mg/dL
13. Macroalbuminuria (urinary albumin excretion rate >300 mg/24h)
14. Baseline Hb <10.5 gm/dL in women, or <13 gm/dL in men
15. Baseline LFT's outside of normal range with the exception of Gilberts Syndrome. (An initial LFT test panel with any values >1.5 times upper limits of normal will exclude a patient; a re-test for any values between normal and 1.5 times normal should be made, and if the values remain elevated above normal limits, the patient will be excluded.)
16. Presence of gallstones (subjects may be eligible two weeks after a laparoscopic cholecystectomy)
17. Portal hypertension, detected by baseline duplex ultrasonography (assessment of direction of flow in right, left and main portal vein [antegrade (normal) or retrograde (abnormal indicative of portal hypertension)]; hemangioma in liver on baseline ultrasonography
18. Untreated proliferative retinopathy
19. Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast-feeding
20. Evidence of sensitization on PRA (determined by demonstration of positive results for anti-HLA antibodies using solid phase immunoassay with soluble HLA Class I molecules as a target, or a general PRA panel with reactivity >20%)
21. Insulin requirement >0.7 IU/kg/day
22. HbA1C >12%
23. Inability to reach the study hospital for transplantation within 24 hrs of notification
24. Untreated hyperlipidemia (fasting LDL cholesterol >130 mg/dL and/or fasting triglycerides >200 mg/dL)
25. Treated hyperlipidemia that is uncontrolled (fasting LDL cholesterol >130 mg/dL; and/or fasting triglycerides >200 mg/dL)
26. Under treatment for a medical condition requiring chronic use of steroids aa. Use of coumadin or other anticoagulant therapy (except aspirin) or subject with PT/INR >1.5

    27. Addison's disease. All subjects should be screened with a basal 8:00 a.m. cortisol test. Results less than the lower limit of normal indicate further testing (e.g., a Cortrosyn stimulation test) to rule out adrenal insufficiency. Abnormal ACTH stimulation test will be an exclusion criterion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2003-08-01 (Actual); Primary Completion 2007-10-23 (Actual); Study Completion 2010-06-24 (Actual)

PRIMARY OUTCOMES:
Insulin independence 12 months after final islet infusion

SECONDARY OUTCOMES:
Basal c-peptide level
Hemoglobin A1c level
Glucose tolerance
C-peptide response to arginine
Mean Amplitude of Glucose Excursion (MAGE)
Mixed meal test

CONTACTS AND LOCATIONS:
Overall Officials: Meredith J Aull, Pharm.D., Principal Investigator — New York Presbyterian Hospital - Weill Cornell Medical Center
Locations (1):
- New York Presbyterian Hospital - Weill Cornell Medical Center, New York, New York, United States